CLINICAL TRIAL: NCT06232915
Title: Accuracy of the Set Tidal Volume During Intraoperative Mechanical Ventilation
Status: Withdrawn | Type: Observational
Why Stopped: Changed to an invitro study using a mechanical lung rather than human subjects.
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chief, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00003946
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Surgery; Mechanical Ventilation Pressure High
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical ventilation: Children requiring mechanical ventilation during a surgical procedure.
  Interventions: Procedure: Mechanical ventilation

INTERVENTIONS:
Procedure: Mechanical ventilation — Mechanical ventilation during surgery

SUMMARY:
Prior to surgery the anesthesia team will be putting a breathing tube into the patient's windpipe and attaching it to a mechanical ventilator (breathing machine). This is to provide oxygen and anesthetic gas, and to help the child breathe while they're asleep. The ventilator also controls the amount of air that moves in and out of the lungs with each breath. This is called tidal volume and that amount is programmed into the machine by the anesthesia team. All of this is standard of care.

As part of the study the investigators will put a small flow sensor between the patient's breathing tube and the tubing from the ventilator. This will measure the amount of air that is moving in and out of the breathing tube. The study team will record the tidal volume that is set on the ventilator and compare it to the airflow measured by the ventilator and the airflow measured by the sensor and see if there is a difference.

ELIGIBILITY:
Inclusion Criteria:

* children aged 0-18 years having surgery at Nationwide Children's Hospital, in whom a cuffed ETT and mechanical ventilation will be used

Exclusion Criteria:

* children with preexisting airway anomalies or respiratory compromise will be excluded from the study.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children requiring intraoperative mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean inspired tidal volume | Baseline
  The average volume of air moved into the lungs over 25 breaths.
Mean expired tidal volume | Baseline
  The average volume of air moved out of the lungs over 25 breaths.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided